CLINICAL TRIAL: NCT01930526
Title: Single Leg Cycling in COPD: Knowledge Translation to Pulmonary Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Principal Investigator, Roger Goldstein, Respirologist, West Park Healthcare Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JREB2011-12
Record Dates: First submitted 2013-07-15; First posted 2013-08-29 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Exercise; Cycling; Single leg; Pulmonary Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pulmonary Rehabilitation (Experimental): Patients will undergo the usual pulmonary rehabilitation programme but instead of two-legged cycling they will undergo single leg cycling where they cycle with one leg for 10-15mins and then the other in the same session.
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Pulmonary Rehabilitation — Pulmonary Rehabilitation (PR) is a short course 6-12 weeks of supervised exercise training and education for patients with COPD. This is part of their usual treatment. This study is replacing two-legged cycling with single leg training. Patients will have the usual PR outcome measures assessed but in addition will have a laboratory exercise test.

SUMMARY:
Pulmonary rehabilitation (PR) with supervised exercise training is a key part of care for patients with chronic lung disease (COPD). Patients can improve their shortness of breath, walking distance and quality of life. However, many patients do not improve their overall fitness. They are too breathless to train at a high enough intensity. In a laboratory training study, patients with COPD improved their overall fitness by using single leg cycling. Despite this knowledge, single leg cycling has not been used clinically. The objective of this project is to use and assess single leg cycling in a clinical setting. Single leg cycling can be incorporated into a clinical service (replacing traditional two legged cycling) as the predominant aerobic training strategy, resulting in improvements in cardio-respiratory fitness (peak oxygen uptake).

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD referred for Pulmonary Rehabilitation

Exclusion Criteria:

* Unstable cardiac disease
* any neurological or orthopaedic condition that would make cycling difficult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in peak oxygen uptake achieved by incremental cycle ergometry | Measured at the end of an average of eight weeks of pulmonary rehabilitation compared to baseline
  A full incremental cardiopulmonary exercise test will be performed on a cycle ergometer to symptom limitation with expiratory gas analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Roger S Goldstein, MBChB, Principal Investigator — West Park Healthcare Centre
Locations (1):
- West Park Healthcare Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Evans RA, Dolmage TE, Mangovski-Alzamora S, Romano J, O'Brien L, Brooks D, Goldstein RS. One-Legged Cycle Training for Chronic Obstructive Pulmonary Disease. A Pragmatic Study of Implementation to Pulmonary Rehabilitation. Ann Am Thorac Soc. 2015 Oct;12(10):1490-7. doi: 10.1513/AnnalsATS.201504-231OC. PMID 26291542